CLINICAL TRIAL: NCT06624774
Title: The Effect of Prehabilitation on Appendicular Skeletal Muscle Mass in Cardiac Patients Awaiting First Time Elective Surgery
Brief Title: Prehabilitation's Effect on Skeletal Muscle Mass in Cardiac Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Stefan Birkett, Chief Investigator, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56646
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
Keywords: prehabilitation; homebased; CABG
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Pilot randomised clinical trial with two groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be partially blinded. The participants in both groups will be blinded from the goal of the measurements taking place. For example, the participants will not be informed specific goal of change of appendicular skeletal muscle mass. The reason for this is, if the participant knows the exact aims of the study, there would be an increased risk of the participants implementing unnatural daily habits, potentially skewing the results. The study cannot be fully blinded due to the exercise and education intervention taking place
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): This group will receive NHS standard care. This includes the 'your heart surgery' - a new beginning booklet at the pre-op assessment 2-4 weeks, before surgery as part of routine care. The leaflet will include information regarding heart procedures, recovery, post-surgery rehabilitation, cardiovascular risk factors, lifestyle advice and support
- Prehabilitation (Active Comparator): Participants randomised to the exercise and education intervention will follow an individualised structured exercise programme and receive group education sessions.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — The structured exercise sessions will be conducted in a homebased setting, consisting of 8 resistance exercises (RE). The 8 RE's will include 4 upper body and 4 lower body exercises (Sit to stand, chest press, heel raises, bicep curls, leg abduction, tricep kickbacks, lunges, mid row). This is adapted from an existing home-based trial in cardiac patients. In addition, the structured exercise programme will include a walking programme. Participants will receive a Fitbit charge 5 activity monitor. Additionally, participants will conduct daily IMT via a Powerbreathe medic plus device. Participants will conduct 6 sets of 6 breaths at 50% of peak inspiratory pressure that has been measured at baseline. Education will be delivered via pre-recorded videos or in person
  Arms: Prehabilitation

SUMMARY:
The study will investigate the effect prehabilitation on skeletal muscle mass via a scanner.

DETAILED DESCRIPTION:
Post COVID 19 data demonstrates vast increases regarding wait times for elective cardiac procedures (104 days). Extended wait times will therefore increase sedentary behaviours, increasing the risk of patient deterioration pre-operatively. Frailty and low muscle mass correlates with poor post-operative outcomes, lower physical function, and lower quality of life. Research regarding prehabilitation in cancer patients demonstrates positive outcomes. Additionally, early research in cardiac patients shows encouraging findings, however, there are limited studies regarding prehabilitation in this cohort of patient. A recent large public, patient involvement (PPI) study was conducted to address the research needs for cardiac patients, carers and medical professionals. Research concerning pre-operative interventions and lifestyle advice where key topics ranking in the top three at the conclusion of the study. Further emphasising the need for studies focusing on prehabilitation. This coupled with no study has assessed the effect of prehabilitation on skeletal muscle provides an important gap in the research to explore.

STUDY SETTING This randomised controlled pilot study will take place at the participant's home and surrounding areas. Data collection will take place at Manchester Metropolitan University.

Patient identification Participants who are cleared for elective surgery and who meet the eligibility criteria will be identified by the surgical team at Manchester University NHS Foundation Trust (Wythenshawe hospital). The investigators will purposively sample individuals from socio-economic deprived areas, ethnic minority backgrounds.

Consent Once identified the surgical team will provide a brief overview of the study and give the potential participant a participant information sheet (PIS). If happy, a consent to be contacted form will be completed by the potential participant. This will be documented in the patient's medical notes by the surgical team. The surgical team will then scan and transfer the completed consent to be contacted document via dropbox for business and a member of the research team will then contact the patient and answer any questions regarding the PIS and study. The potential participants will have 72hrs to decide if they want to take part in the study. If the potential participant has not decided after 72hrs, they will be able to contact the research team for the next 5 working days, if they have decided they want to participate. For those who decide to take part, written consent will be obtained at their baseline assessment.

Withdrawal Criteria Participants will be informed that they are able to withdraw from the study at any time. The chief investigator has the right to withdraw the participant from the trial if appropriate, for example if the participants circumstances have changed since the start of the study. The reasons for withdrawal will be recorded.

Randomisation- Method of implementing the allocation sequence Participants will be randomised in a 1:1 ratio via sealed envelope (https://www.sealedenvelope.com), a secure computerised randomisation programme. Sealed envelope will maintain the allocation sequence concealment, only the participant study number will be entered into the system.

ELIGIBILITY:
Inclusion Criteria:

* • Between the age of 18-85.

  * First time elective cardiac surgery patients who have been deemed clinically stable by the surgical team.
  * Able to speak and understand English.
  * Medically optimised.
  * Absence of contraindications to exercise and exercise testing following the guidance of the Association of Chartered Physiotherapist in Cardiovascular Rehabilitation (ACPICR) and British Association of Cardiovascular Prevention and Rehabilitation (BACPR).

Exclusion Criteria:

* • Patients with coexisting congenital heart conditions, significant comorbidities including heart failure (left ventricular ejection fraction (LVEF) <35%), advanced cancer and conditions preventing the patient from providing informed consent.

  * Patients with open wounds, ongoing complications and systemic infections
  * Contraindications to inspiratory muscle training (Severe asthma exacerbations, recently perforated ear drum, large bullae, history of spontaneous pneumothorax). Following guidance from a recent prehabilitation randomised controlled trial (19).
  * Recent thoracic surgery (< 1 year).
  * Individuals who do not understand English or have a disability that limits their capacity to understand verbal explanations.
  * Those who are currently involved in other research studies.
  * Women who are pregnant or breastfeeding.
  * Current drug abusers and excessive alcohol drinkers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study will be the change in appendicular skeletal muscle mass (KG/M2). | Baseline, 12 weeks and one week prior to surgery
  Appendicular skeletal muscle mass will be measured via DEXA scan

SECONDARY OUTCOMES:
Pre-operative preparedness for surgery | recorded one-week pre operation
  Participants will conduct a pre-operative preparedness for surgery questionnaire adapted from Kenton, Pham (32). The questionnaire will consist of 10 questions, regarding the surgical procedure and surgical aftermath
Handgrip strength | Baseline, 12 weeks and one week prior to surgery
  Hand grip assessment will be performed by hand dynamometer (JAMAR plus) and the method used will be the Southampton protocol. Participants will squeeze the hand dynamometer for 5 seconds. This will be performed three times by each arm with the highest score being recorded
Physical Performance | Baseline, 12 weeks and one week prior to surgery
  The SPPB will is a validated method to assess physical function (25). The test will consist of three timed tasks that assess the patients gait speed, standing balance and chair sit to stand. Individual scores are given for each test based on the defined cut-off points. The score then be calculated with 0 being the lowest score and 12 being the highest
Aerobic capacity | Baseline, 12 weeks and one week prior to surgery
  Via a six minute walk self paced test
Health related Quality of Life | Baseline, 12 weeks and one week prior to surgery
  Quality of life will be obtained via a 5-component scale questionnaire (EQ-5D-5L). The questionnaire will measure mobility, self-care, usual activities, pain/discomfort and anxiety and depression. Additionally, the questionnaire will include a 20cm analogue scale labelled from 0-100 aimed to assess patient health on the day, 100 will corelate with the best health possible and 0 will align with the worst
Inspiratory muscle function | Baseline, 12 weeks and one week prior to surgery
  Maximal inspiratory pressure will be conducted to assess inspiratory muscle strength utilising a handheld respiratory pressure meter. The same pressure gauge will be used for all testing and calibrated to certify accuracy. Each participant will perform the manoeuvre 5 times, the aim is to have the two highest values within 10cmH20
Anxiety and depression | Baseline, 12 weeks and one week prior to surgery
  Anxiety and depression will be measured via the Hospital anxiety and depression questionnaire (HADS). The questionnaire will be presented in the form of a 0-3 Likert scale. Participants will have a total of 14 questions to answer, 7 anxiety questions and 7 depression questions
Nutrition | Baseline, 12 weeks and one week prior to surgery
  Participants will conduct a 5-day food diary via the digital application Libro. This will allow for the measurements of total calories (Kcals), protein intake, fat intake and carbohydrate intake
Adherence | Baseline, 12 weeks and one week prior to surgery
  Adherence will be assessed by monitoring participant logbook entries to account for participant adherence to exercise protocol, during the study. Entries will include, completed exercise sessions and partially completed sessions. Drop-out from the programme will also be documented for both study groups in addition to the reasons for drop-out, where provided by the participants
Blood Pressure | Baseline, 12 weeks and one week prior to surgery
  Blood pressure will be measured via the Omron blood pressure monitor (Omron Healthcare, Milton Keynes, United Kingdom).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Birkett, PhD, Principal Investigator — Manchester Metropolitan University
Locations (1):
- Manchester University NHS Foundation Trust, Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers outside of this project.